CLINICAL TRIAL: NCT04634292
Title: Processus Attentionnels impliqués Dans la Locomotion Chez l'Enfant à développement Typique et l'Enfant Atteint de Paralysie cérébrale : Une étude EEG.
Brief Title: Dual Tasking in Children With Cerebral Palsy and Healthy Children: an EEG Study
Acronym: PRALOC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.067; 2020-A00470-39 (Other: ID RCB)
Record Dates: First submitted 2020-09-03; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children with cerebral palsy 7-9 years: 21 children
  Interventions: Behavioral: EEG
- Children with cerebral palsy 10-12 years: 21 children
  Interventions: Behavioral: EEG
- Healthy children 7-9 years: 21 children
  Interventions: Behavioral: EEG
- Healthy children 10-12 years: 21 children
  Interventions: Behavioral: EEG

INTERVENTIONS:
Behavioral: EEG — EEG + walking task + auditory task

SUMMARY:
Simultaneous execution of motor and cognitive tasks is embedded in the daily life of children. An EEG study will be conducted on healthy children and children with cerebral palsy to study the neural correlates during dual tasking while walking

DETAILED DESCRIPTION:
Children will walk at their preferred speed on a treadmill. During dual tasking, they will listen to animals cries and will have to count the number of specified animals cries.

ELIGIBILITY:
Inclusion Criteria:

* normal walking

For children with cerebral palsy: diplegia or hemiplegia, GMFCS 1 or 2, no botulinium injection since 4 months

Exclusion Criteria:

* medical problem

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children and children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Neural correlates during dual tasking in children | 2 years
  EEG, locomotion parameters, cognitive performances

IPD SHARING:
Plan to Share IPD: Undecided